CLINICAL TRIAL: NCT06535464
Title: Hypotension Prediction Index (HPI) in Patients Undergoing Robotic Assisted Radical Prostatectomy
Acronym: HPI in RARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, Prof, University of Foggia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 135/C.E. 2021
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Hypotension During Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed therapy guided by Hypotension Prediction Index algorithm (Active Comparator)
  Interventions: Device: Hypotension Prediction Index
- Goal-directed therapy alone (Sham Comparator)
  Interventions: Device: No Hypotension Prediction Index

INTERVENTIONS:
Device: Hypotension Prediction Index — Fluid management guided by Hypotension Prediction Index
  Arms: Goal-directed therapy guided by Hypotension Prediction Index algorithm
Device: No Hypotension Prediction Index — Fluid management not guided by Hypotension Prediction Index
  Arms: Goal-directed therapy alone

SUMMARY:
Robot assisted radical prostatectomy (RARP) is the leader in robotic treatment for prostate cancer. Goal-directed therapy (GDT) is the approach used, but HPI, a machine learning algorithm analysing arterial waveforms, might offer additional benefits. The aim of this prospective randomised study is to evaluate the cumulative amount of intraoperative arterial hypotension episodes in patients undergoing RARP managed by GDT protocol guided or not by HPI algorithm

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients undergoing RARP; American Society of Anaesthesiology (ASA) SCORE I-III

Exclusion Criteria:

* Body Mass Index (BMI) of 18.5 to 35, uncontrolled arrhythmias, myocardial infarction or ischemic/hemorrhagic stroke in the last 6 months, III/IV stage Global Initiative for Chronic Obstructive Lung Disease, pulmonary fibrosis, contraindication to radial artery cannulation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
cumulative amount of time spent in Hypotension | intraoperative
  the cumulative amount of intraoperative hypotension, measured by Time Weighted Average (TWA) of Mean Arterial Pressure (MAP) below 65 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedali Riuniti, Foggia, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No
It is not allowed in the consent form

REFERENCES:
- [Derived] Cotoia A, Discenza A, Rauseo M, Matella M, Caggianelli G, Ciaramelletti R, Mirabella L, Cinnella G. Intraoperative hypotension during robotic-assisted radical prostatectomy: A randomised controlled trial comparing standard goal-directed fluid therapy with hypotension prediction index-guided goal-directed fluid therapy. Eur J Anaesthesiol. 2025 Oct 1;42(10):916-923. doi: 10.1097/EJA.0000000000002211. Epub 2025 Jun 9. PMID 40493027